CLINICAL TRIAL: NCT03895996
Title: A Phase 1 / 2 Double-Blind, Randomized, Placebo Controlled Study of Safety, Tolerability and Potential Efficacy of AVOTRES Cell-Based Therapy (AVT001) in Patients With Type 1 Diabetes
Brief Title: Safety, Tolerability and Potential Efficacy of AVT001 in Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Avotres Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVT001-T1D-01
Record Dates: First submitted 2019-03-15; First posted 2019-03-29 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AVT001 (Treatment) (Experimental): Infusion of AVT001 (treatment)
  Interventions: Drug: AVT001
- Matched placebo (Placebo Comparator): Infusion of AVT001-matched placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AVT001 — autologous dendritic cell therapy
  Arms: AVT001 (Treatment)
Other: Placebo — matched placebo
  Arms: Matched placebo

SUMMARY:
This is a double-blind, randomized , placebo-controlled study to evaluate the safety and tolerability of AVT001, and to assess AVT001 as a potential treatment for type 1 diabetes (T1D). The trial will involve approximately 24 new-onset T1D subjects.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of type 1 diabetes, within 12 months of first dosing, confirmed by positive lab result for one or more of the following types of autoantibodies:

   1. Glutamic acid decarboxylase (GAD65)
   2. Insulinoma associated protein 2 (IA-2, also known as ICA-512)
   3. Zinc transporter 8 (ZnT8).
2. Age 16 or older and able to provide informed consent/assent.
3. If a participant is female with reproductive potential, willing to avoid pregnancy through the duration of the trial.
4. Signed and dated written informed consent/assent.

Key Exclusion Criteria:

1. Poorly controlled diabetes despite insulin therapy, who in the opinion of the investigator would not be a good candidate for participation in a clinical trial
2. Screening hemoglobin <10.0 g/dL; leukocytes <3,000/uL; neutrophils <1,500/uL; lymphocytes <800/uL; platelets <100,000/uL
3. Screening Urine Albumin Excretion > 300mg/gmCr
4. Screening eGFR < 60 mL/min/1.73m2
5. Screening ALT or AST > 1.5x upper limit of normal (ULN)
6. Screening bilirubin > 2.0 mg / dL, or > 3.0 mg / dL for participants with Gilbert's Syndrome
7. Current use of immunosuppressive or immunomodulatory therapies, including pharmacologic doses of systemic steroids. However, topical steroidal creams and inhaled steroids without large systemic absorption are allowed.
8. Coincident medical condition likely to require immunosuppressive or immunomodulatory therapies.
9. Coincident medical condition likely to limit short term (5 year) life expectancy (malignancy, symptomatic coronary artery disease, recent stroke)
10. Prior radiation therapy, immunotherapy (within 1 year of screening), or chemotherapy
11. Serologic evidence of current HIV-1 or HIV-2 infection
12. Serologic evidence of hepatitis C infection
13. Serologic evidence of acute or chronic active hepatitis B as measured by Core Ab positive and / or Surface Antibody antigen positive
14. Subjects with other autoimmune conditions (except compensated or treated autoimmune thyroid, celiac, alopecia, or vitiligo diseases)
15. Women who are pregnant (pregnancy testing during screening), breastfeeding, or planning pregnancy during the study period
16. Inadequate venous access to support leukapheresis
17. Any condition that in the opinion of the investigator(s) would preclude the subject from participating in a clinical trial.
18. Abnormal screening ECG that in the opinion of the investigator or sponsor would pose a safety risk.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2023-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gaglia, MD, Principal Investigator — Joslin Diabetes Center, Harvard Medical School
Locations (1):
- Joslin Diabetes Center, Harvard Medical School, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gaglia JL, Daley HL, Bryant NK, Ritz J, Dong T, Skyler JS, Jiang H. Novel Autologous Dendritic Cell Therapy AVT001 for Type 1 Diabetes. NEJM Evid. 2024 Jul;3(7):EVIDoa2300238. doi: 10.1056/EVIDoa2300238. Epub 2024 Jun 25. PMID 38916421
- See also: Avotres Inc. in collaboration with Joslin Diabetes Center, a Harvard Medical School affiliate, have reported one year data of a phase I/II clinical trial of AVT001 in type 1 diabetes. — https://www.einpresswire.com/article/722881487/avt001-phase-i-ii-clinical-trial-1-year-data-in-type-1-diabetes-is-published

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AVT001 (Treatment) | Matched Placebo
Started | 16 | 9
Leukapheresed and Dosed | 16 | 9
Primary Analysis at Day 150 | 16 | 9
Supplemental Analysis at Day 360 | 16 | 8
Completed | 16 | 8
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AVT001 (Treatment) | Matched Placebo | Total
Number analyzed (Participants) | 16 | 9 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (9.0) | 26.2 (6.2) | 26.4 (8.0)
Age, Customized [Count of Participants; unit: Participants]
  Age by Category: <18 | 2 | 1 | 3
  Age by Category: 18-<25 | 7 | 4 | 11
  Age by Category: 25-<40 | 6 | 4 | 10
  Age by Category: 40-<60 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 10 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 13 | 9 | 22
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Description: Treatment-emergent AEs (TEAEs) are defined as any AE that started on or after the first dose of study medication through 30 days following the last dose.
Time Frame: At the Primary Analysis (when all the patients have completed their Day 150 visit)
Population: The safety (SAF) population is defined as all subjects who receive at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | AVT001 (Treatment) | Matched Placebo
Number analyzed (Participants) | 16 | 9
participants
  Participants with Any TEAE | 9 | 6
  Neutrophil count decreased | 4 | 1
  Hyponatraemia | 3 | 1
  Cough | 3 | 0
  White blood cell count decreased | 2 | 1
  Ear pain | 2 | 0
  Lymphocyte count decreased | 2 | 0
  Dizziness | 1 | 2
  Anaemia | 1 | 1
  Blood bicarbonate decreased | 1 | 1
  Blood bilirubin increased | 1 | 1
  Corona virus infection | 1 | 1
  Fatigue | 1 | 1
  Hypocalcaemia | 1 | 1
  Pyrexia | 1 | 1
  Chills | 1 | 0
  Gastrooesophageal reflux disease | 1 | 0
  Joint dislocation | 1 | 0
  Nasal congestion | 1 | 0
  Non-cardiac chest pain | 1 | 0
  Oropharyngeal pain | 1 | 0
  Palpitations | 1 | 0
  Sinusitis | 1 | 0
  Headache | 0 | 2
  Blood potassium decreased | 0 | 1
  Gastroenteritis | 0 | 1
  Influenza like illness | 0 | 1
  Nausea | 0 | 1
  Oral papule | 0 | 1
  Upper-airway cough syndrome | 0 | 1

2. Primary Outcome: Number of Participants and Severity of Local i.v.-Site Reactions,
Description: Number of Participants and severity of local intravenous site reactions after receiving the three doses are reported.
Time Frame: 5 months post first dose
Population: The safety (SAF) population is defined as all subjects who receive at least one dose of study medication.
Measure: Number; unit: Number of patients
Arm/Group | AVT001 (Treatment) | Matched Placebo
Number analyzed (Participants) | 16 | 9
Number of patients | 0 | 0

3. Primary Outcome: Changes From Baseline of Creatinine
Description: Safety/tolerability outcomes - creatinine
Time Frame: 5 months post first dose
Population: The safety (SAF) population is defined as all subjects who receive at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | AVT001 (Treatment) | Matched Placebo
Number analyzed (Participants) | 16 | 9
umol/L | 1.9338 (7.51638) | 0.4911 (5.48705)

4. Primary Outcome: Changes From Baseline of Aspartate Aminotransferase
Description: Safety/tolerability outcomes - Aspartate Aminotransferase
Time Frame: 5 months post first dose
Population: The safety (SAF) population is defined as all subjects who receive at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | AVT001 (Treatment) | Matched Placebo
Number analyzed (Participants) | 16 | 9
U/L | -1.9 (7.76) | 2.2 (6.10)

5. Primary Outcome: Changes From Baseline of Alanine Aminotransferase
Description: Safety/tolerability outcomes - Alanine Aminotransferase
Time Frame: 5 months post first dose
Population: The safety (SAF) population is defined as all subjects who receive at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | AVT001 (Treatment) | Matched Placebo
Number analyzed (Participants) | 16 | 9
U/L | -0.1 (5.21) | 1.1 (3.26)

6. Primary Outcome: Changes From Baseline of Total Bilirubin
Description: Safety/tolerability outcomes - Total Bilirubin
Time Frame: 5 months post first dose
Population: The safety (SAF) population is defined as all subjects who receive at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | AVT001 (Treatment) | Matched Placebo
Number analyzed (Participants) | 16 | 9
umol/L | -0.114 (4.0603) | 0.000 (4.0103)

7. Secondary Outcome: Assessment of the HLA-E-restricted CD8+ T Cell Regulatory Activity ("Potency Assay")
Description: CD8+ T cell Inhibition Assay is used to determine whether AVT001 corrects the defect of the dysfunctional Q/E CD8+ Treg pathway in T1D patients. More specifically, this assay detects the specific recognition between the TCR on patients' Q/E CD8+Treg cells and the "common target structure", the HLA-E/Hsp60sp complex, expressed on the surface of the artificially established target cells.
  The % inhibition measures the function of down-regulation by Q/E CD8+ Tregs via comparing the % of inhibition of TH1 cells versus TB1 cells.
  By assessing the % inhibition of the TH1 cells of the patient's CD8+ T cells, the CD8+ T cell Inhibition Assay detects the specific recognition of the common target structure (HLA-E/Hsp60sp) on TH1 cells by the TCR on the patient's T cells to be tested.
  A negative value means the measured Q/E CD8+ Tregs completely lose its inhibition function, and the TH1 cells cultured with it happened to grow faster than the corresponding TB1 cells as its control.
Time Frame: 5 months post first dose
Population: The pharmacodynamic (PD) population is defined as all subjects in the safety population with at least one post-baseline assessment for the evaluation of the CD8+ T-cell reg system biomarker.
Measure: Mean (Standard Deviation); unit: Percent of Inhibition
Arm/Group | AVT001 (Treatment) | Matched Placebo
Number analyzed (Participants) | 16 | 9
Percent of Inhibition
  Baseline | -11.2 (9.9) | 3.5 (7.1)
  Visit Day 150 | 9.3 (24.9) | 1.8 (15.1)

8. Secondary Outcome: Changes From Baseline in the Area Under the Curve (AUC) of the Stimulated C-peptide Levels Over a 4-hour Mixed Meal Tolerance Test (MMTT)
Description: The area under the stimulated C-peptide curve (AUC) over the first 4-hour period of a mixed meal glucose tolerance test is calculated using the trapezoidal rule that is a weighted sum of the C-peptide values over the 240 minutes. The AUC is normalized by dividing it with 240 mins, therefore, its unit is nmol/L. Missing C-peptide levels at any given timepoint is not imputed. In the calculation of the AUC when C-peptide levels are missing, a line is drawn from the last timepoint with a non-missing C-peptide to the next timepoint with non-missing C-peptide.
Time Frame: 5 months post first dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | AVT001 (Treatment) | Matched Placebo
Number analyzed (Participants) | 16 | 9
nmol/L
  Baseline | 0.531 (0.3628) | 0.611 (0.1776)
  Visit Day 150 | 0.518 (0.4299) | 0.472 (0.1342)

9. Secondary Outcome: Changes From Baseline in HbA1c
Description: HbA1c is a blood test that is used to monitor blood glucose control in people with diabetes.
  HbA1c is short for glycated haemoglobin. The test is also sometimes called haemoglobin A1c.
Time Frame: 5 months post first dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % of glycated haemoglobin in the blood
Arm/Group | AVT001 (Treatment) | Matched Placebo
Number analyzed (Participants) | 16 | 9
% of glycated haemoglobin in the blood
  Baseline | 6.0375 (0.73201) | 5.6556 (0.67289)
  Visit Day 150 | 6.1500 (0.84538) | 5.8222 (0.84080)

ADVERSE EVENTS:
Time Frame: All anticipated and unanticipated adverse events occured during the study (2 years), including both Treatment Emergent Adverse Events (TEAEs) and Post-Treatment Adverse Events (PTAEs), that exceed a 5% frequency threshold within any arm of the clinical study.
Description: No difference from the clinicaltrials.gov definitions. There has been no death or SAE events recorded throughout the study, and therefore 0 was reported in the following table.
Arm/Group | AVT001 (Treatment) | Matched Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/9
Other Adverse Events (participants affected / at risk) | 16/16 | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AVT001 (Treatment) (N=16) | Matched Placebo (N=9)
White blood cell count decreased (Investigations) | 7 | 5
Blood bicarbonate decreased (Investigations) | 6 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 1
Corona virus infection (Infections and infestations) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 2
Neutrophil count decreased (Investigations) | 4 | 3
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1
Lymphocyte count decreased (Investigations) | 3 | 0
Blood bilirubin increased (Investigations) | 2 | 4
Ear pain (Ear and labyrinth disorders) | 2 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Pyrexia (General disorders) | 2 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Fatigue (General disorders) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Gastrooesophageal reflux disease (General disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Monocyte count decreased (Investigations) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oral papule (Gastrointestinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT03895996/Prot_SAP_000.pdf